CLINICAL TRIAL: NCT02012751
Title: Nevus Doctor Clinical Decision Support Program for Pigmented Skin Lesions and Melanoma
Brief Title: Nevus Doctor Clinical Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1206
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-06

CONDITIONS: Nevus; Melanoma
Keywords: Computer-assisted diagnosis; General practice; Dermatoscopy; Melanoma; Nevus
MeSH Terms: conditions — Nevus; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nevus doctor program (Experimental): Use of Nevus doctor program to assess the diagnostic category of pigmented skin lesions
  Interventions: Device: Nevus doctor program

INTERVENTIONS:
Device: Nevus doctor program — The Nevus doctor program supplies a diagnostic category of pigmented skin lesions based on dermatoscopy images.

SUMMARY:
The "Nevus doctor" is a dermatoscopy based computer decision support tool to assist general practitioners (GPs) in the classification of pigmented skin lesions (PSLs). The aim of the program "Nevus doctor" is to help GPs increase their diagnostic accuracy, in particular regarding the selection of suspicious PSLs that need biopsy or referral to specialist health care for further assessment. The aim of this study is to investigate the diagnostic performance of the decision support tool in a primary care setting in Norway. We hypothesize that the diagnostic accuracy of the computer program "Nevus doctor" is better than the performance of the GPs.

DETAILED DESCRIPTION:
In the trial GPs examine patients who attend a primary health care center. A given PSL is first assessed clinically by the GP and afterwards photographed. A clinical photograph as well as a dermatoscopic photograph is taken, the latter using a dermatoscope attached to the lens of the camera. The dermatoscopic image is then processed by the computer program. The performance of "Nevus doctor" is compared with the GPs' assessment. A dermatologist reviews all cases based on the clinical and dermatoscopic photographs and this assessment serves as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Pigmented skin lesion

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of correct test results | Up to 2 weeks from enrollment
  The computer program tests whether the appearance of a skin lesion is suggestive of skin cancer. There are two possible test outcomes: "suspicious" or "not suspicious". The reference standard is the assessment done by a dermatologist. The number (and percentage) of skin lesions correctly classified as "suspicious" or "not suspicious" is reported. Furthermore sensitivity, specificity, positive and negative predictive values are calculated.

SECONDARY OUTCOMES:
Patterns regarding false test results | Up to 2 weeks from enrollment
  All cases with false test results are described in order to identify any pattern that can help to explain the false test result: correlation with specific types of skin lesions, poor image quality, gender and age of the patients.

OTHER OUTCOMES:
User-friendliness | 6-8 months after enrollment
  Participating GPs are invited to interviews

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Schopf, Ph.D., Principal Investigator — University Hospital North-Norway
Locations (1):
- Kirkenes Legesenter, Kirkenes, Finnmark Fylke, Norway